CLINICAL TRIAL: NCT00002118
Title: An Open-Label Safety Program for the Use of Zalcitabine (Dideoxycytidine; ddC) in Pediatric Patients With Symptomatic HIV Infection Who Have Failed or Are Intolerant to AZT Monotherapy, or Who Have Completed Other ddC Protocols, or Are Ineligible for Other Ongoing Clinical Studies
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Organization: NIH AIDS Clinical Trials Information Service (Industry)
Masking: None | Purpose: Treatment
Other Study IDs: 031F; NV14610
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 1997-08

CONDITIONS: HIV Infections
Keywords: Zalcitabine; Acquired Immunodeficiency Syndrome; AIDS-Related Complex
MeSH Terms: conditions — HIV Infections; Acquired Immunodeficiency Syndrome; AIDS-Related Complex | interventions — Zalcitabine

INTERVENTIONS:
Drug: Zalcitabine

SUMMARY:
To allow, on a compassionate use basis, zalcitabine (ddC) for pediatric patients with symptomatic HIV disease who have failed treatment or who are intolerant to zidovudine (AZT), or who have completed other ddC protocols, or who are ineligible for ongoing clinical trials.

DETAILED DESCRIPTION:
Patients receive ddC and are evaluated at study entry and every 3 months thereafter, until 3 months after ddC becomes approved for pediatric patients or the sponsor deems it necessary to terminate the protocol.

ELIGIBILITY:
Inclusion Criteria

Patients must have:

* Symptomatic HIV infection.
* Failure on or intolerance to AZT monotherapy OR completed other ddC protocols OR been ineligible for other ongoing clinical trials.
* Consent of parent or guardian required.

Note:

* Patients who do not meet the eligibility requirements may discuss their cases with the medical monitor.

Ages: 3 Months to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 600

CONTACTS AND LOCATIONS:
Locations (1):
- Hoffmann - La Roche Inc, Nutley, New Jersey, United States

REFERENCES:
- [Background] Adkins JC, Peters DH, Faulds D. Zalcitabine. An update of its pharmacodynamic and pharmacokinetic properties and clinical efficacy in the management of HIV infection. Drugs. 1997 Jun;53(6):1054-80. doi: 10.2165/00003495-199753060-00009. PMID 9179531